CLINICAL TRIAL: NCT05240820
Title: Clinical Outcomes Associated With the Use of Polyglactin 910 (Vicryl®) and Polypropylene (Prolene®) Suture, and Polydioxanone (StratafixTM Spiral PDS® Plus) and Combination of 2-Octyl Cyanoacrylate and Polyester Mesh (Dermabond Prineo®) for Multi-Layer Wound Closure Following Excision of Giant Benign Tumors
Brief Title: A Comparative Study of Scar Quality and Safety According to Suture Materials Following Excision of Benign Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Johnson and Johnson Medical Korea Ltd (Unknown)
Responsible Party: Principal Investigator, Moon, Kyung Chul, Clinical Assistant Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WC-2020-09
Record Dates: First submitted 2022-02-05; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Scar Quality Assessment and Safety
Keywords: Scar quality; Safety; Suture; Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicryl+Prolene (Placebo Comparator): wound closure using polyglactin 910 (Vicryl®, Ethicon, Johnson and Johnson Ltd., NJ, USA) and polypropylene (Prolene®, Ethicon)
  Interventions: Procedure: multi-layer wound closure
- PDS+Dermabond (Active Comparator): wound closure using polydioxanone (StratafixTM Spiral PDS® Plus) and combination of 2-octyl cyanoacrylate and polyester mesh (Dermabond Prineo®)
  Interventions: Procedure: multi-layer wound closure

INTERVENTIONS:
Procedure: multi-layer wound closure — We prospectively analyze clinical outcome data from 30 subjects who perform multi-layer wound closure using polyglactin 910 and polypropylene, and polydioxanone and combination of 2-octyl cyanoacrylate and polyester mesh following excision of giant benign tumors.

SUMMARY:
Due to the rise in the incidence of giant benign tumors such as lipoma, excision of benign tumors on body have been performed by plastic surgeons. After excision of giant benign tumors, efforts should be include with a goal of achieving optimal cosmetic outcomes after subcutaneous and dermal sutures may be important to improve scar quality because suture methods might influence the final aesthetic outcome. Various absorbable suture materials have been used for tension-relieving deep sutures. Subcutaneous and dermal sutures using Polygalctin 910 (Vicryl®, Ethicon, Johnson and Johnson Ltd.), which is absorbable, synthetic, braided suture composed of a copolymer made from 90% glycolide and 10% L-lactide or polydioxanone (PDS®, Ethicon), which is composed of polyester and p-dioxanone with skin suture using polypropylene (Prolene®, Ethicon) have been commonly used after excision of tumors.

Although these sutures are particularly useful where combination of absorbable suture and extended wound support for up to six weeks is desirable, strong and secure skin sutures may be needed to improve scar quality following excision of tumors on back and abdomen due to their thick skins. However, increased wound closure times are their drawbacks. To overcome these drawbacks, a new subcutaneous suture material composed of polydioxanone, StratafixTM Spiral PDS II® and a new skin suture material using combination of 2-octyl cyanoacrylate and polyester mesh (Dermabond Prineo®, Ethicon) have been developed and skin sutures using combination of these two materials may be an alternative suture method to decrease wound closure times and improve scar quality for better wound closure with high-tension closure, favorable and encouraging results compared to traditional suture methods.

Although polyglactin 910, polydioxanone, polypropylene, and combination of 2-octyl cyanoacrylate and polyester mesh have been used in general surgery and neurosurgery, no studies on the clinical outcomes, specifically on scar quality after excision of tumors have been reported in plastic surgery. Therefore, the purpose of this study is to compare clinical outcomes associated with scar quality between the use of polyglactin 910 and polypropylene suture, and polydioxanone and combination of 2-octyl cyanoacrylate and polyester mesh for multi-layer wound closure following excision of giant benign tumors.

DETAILED DESCRIPTION:
We prospectively analyze clinical outcome data from 30 subjects who perform multi-layer wound closure using polyglactin 910 (Vicryl®, Ethicon, Johnson and Johnson Ltd., NJ, USA) and polypropylene (Prolene®, Ethicon), and polydioxanone (StratafixTM Spiral PDS® Plus) and combination of 2-octyl cyanoacrylate and polyester mesh (Dermabond Prineo®) following excision of giant benign tumors. Patients are randomized into two groups: one sutured by polyglactin 910 and polypropylene and the other group sutured by polydioxanone and combination of 2-octyl cyanoacrylate and polyester mesh. For a group sutured by polyglactin 910 and polypropylene, deep dermal layer will be sutured by polyglactin 910 and polypropylene will be used for suture of superficial dermis and epidermis. For the other group sutured by polydioxanone and combination of 2-octyl cyanoacrylate and polyester mesh, deep dermal layer will be sutured by polydioxanone and polyester mesh will be applied for approximation of superficial dermal layer and epidermis.

A computer-generated list, created using random permuted blocks of 6, that is stratified by hospital will be used for randomization. The allocation configuration will be generated and concealed until interventions will be assigned by a secretary not involved in this trial. Patients with benign tumors greater than 20cm2 (expected scar length more than 3cm) will be included in this study. A Sonography or magnetic resonance imaging scan with millimeter slices will be performed to measure the size of the tumors.

Based on previous studies, the number of subjects was calculated in this study. The weighted scar quality was 2.85 ± 0.57 in one group and 1.96 ± 0.58 in the other group. The following values were used to calculate the number of subjects: Type I error (α) = 5%, power of test = 95%. Independent t-test was used to calculate sample size and differences between two independent means of two groups were used for calculation of sample size. Actual power was 0.954 and the calculation result of the sample size in each group was 10. Considering a drop-out rate of broadly 30%, the number of subjects in each group was 14.3 (=10/(1-0.30)) and a sample size of 30 (=15 × 2) randomly assigned subjects was required.

Differences between the randomized groups will be tested for statistical significance using the Pearson's Chi-Square test for categorical variables. For continuous variables, the independent t-test or Wilkoxon rank-sum test for independent samples will be used for not normally distributed variables. Both intention-to-test (ITT) and per-protocol (PP) analyses will be performed. The median operative time to complete wound closure was also estimated using the Kaplan-Meier method. A P-value < 0.05 is considered statistically significant. All statistical analyses are performed using SPSS for Windows, version 12.0 (SPSS, Inc, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign tumors greater than 20cm2
* Patients with expected scar length (incision length) longer than 3cm
* Patients who need excision of benign tumors

Exclusion Criteria:

* Pregnancy, lactation, patients with previous scars around the benign tumors
* Patients with wound infection, human immunodeficiency virus positive

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-05 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
the Patient and Observer Scar Assessment Scale (POSAS) | six months
  aesthetic outcome as assessed by the overall impression

SECONDARY OUTCOMES:
the Patient and Observer Scar Assessment Scale (POSAS) | three months
  aesthetic outcome as assessed by the overall impression

OTHER OUTCOMES:
Postoperative complications | six months
  suture material exposure, hemorrhage, surgical site infection, wound infection, skin necrosis, wound dehiscence, seroma rates, and hyper- or hypoesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Chul Moon, MD, PhD, Principal Investigator — ICJME

IPD SHARING:
Plan to Share IPD: No